CLINICAL TRIAL: NCT05046600
Title: Multi-Center, Prospective Registry to Evaluate the Continued Safety and Effectiveness of Hand and Wrist Products
Brief Title: Registry of Arthrex Hand and Wrist Products
Status: Recruiting | Type: Observational
Sponsor: Arthrex, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: AIRR-0010
Record Dates: First submitted 2021-08-31; First posted 2021-09-16 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Ulnar/Radial Collateral Ligament Reconstruction; Ligament Repair or Reconstruction; Small Bone Fragments and Arthrodesis; Scapholunate Ligament Reconstruction; Carpal Fusion (Arthrodesis) of the Hand; Digital Tendon Transfers; Carpometacarpal Joint Arthroplasty; Arthrodesis; Digital Tendon Transfer; Distal Radius Fracture Fixation
MeSH Terms: conditions — Ankylosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- All Products listed in Descriptions: Biocomposite™ or PEEK PushLock, DX SwiveLock SL, Headless Compression Screws, Tenodesis Screw (Biocomposite and PEEK), Corkscrew® Titanium (Nano and Micro-Corkscrew), DynaNite Nitinol Staples KreuLock Screws
  Interventions: Device: Products listed in cohort description

INTERVENTIONS:
Device: Products listed in cohort description — Depending on approved indication per product

SUMMARY:
A Multi-Center, Prospective Registry to Evaluate the Continued Safety and Effectiveness of Hand and Wrist Products

DETAILED DESCRIPTION:
The objective of the registry is to evaluate the continued safety and effectiveness of the Arthrex hand and wrist products including the Biocomposite or PEEK PushLock® Anchors for ulnar/radial collateral ligament reconstruction; and/or the DX SwiveLock® SL Anchors (3.5 x 8.5mm) for ligament repair or reconstruction (e.g. scapholunate ligament reconstruction, ulnar/radial collateral ligament reconstruction, and carpometacarpal joint arthroplasty); and/or, the Headless Compression Screws for small bone fragments; and/or, the arthrodesis Tenodesis Screw (Biocomposite and PEEK), for ulnar collateral ligament reconstruction; and/or, the Corkscrew® Titanium Anchor (Micro Corkscrew® Anchor) for ulnar/radial collateral ligament reconstruction, digital tendon transfers (Nano Corkscrew® Anchor); and/or, the DynaNite® Nitinol Staples for carpal fusion (arthrodesis) of the hand; and/or, the KreuLock™ Screws for Distal Radius

ELIGIBILITY:
Inclusion Criteria:

1. Subject requires surgery using Arthrex hand and wrist implants included in the registry.
2. Subject is 18 years of age or over.
3. Subject is not considered a vulnerable subject (i.e. child, pregnant, nursing, prisoner, or ward of the state).
4. Subject signed informed consent and is willing and able to comply with all registry requirements

Exclusion Criteria:

1. Insufficient quantity or quality of bone.
2. Blood supply limitations and previous infections, which may retard healing.
3. Foreign-body sensitivity or foreign-body reactions.
4. Any active infection or blood supply limitations.
5. Conditions that tend to limit the patient's ability or willingness to restrict activities or follow directions during the healing period.
6. Subjects that are skeletally immature -

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Approximately 50 subjects, male and female, 18 years of age or older will be enrolled for each product and material.
  Subjects will be recruited from the surgeon's patient population or referrals from other physicians.
Sampling Method: Non-Probability Sample
Enrollment: 650 (Estimated)
Dates: Start 2021-07-20 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
To assess a change in Visual Analogue Scale (VAS) survey | Preoperatively, 3 months, 6 months and 12 months postoperatively
  Patient reported pain scale 0-10 point scale (0 min,10 max)

SECONDARY OUTCOMES:
To assess a change in Veterans Rand 12-Item Health Survey (VR-12) | Preoperatively, 3 months, 6 months and 12 months postoperatively
  Patient reported changes in general health and mental survey. Average score is 50 (negative answers bring scores down, positive answers bring scores up

OTHER OUTCOMES:
Quick Disabilities of the Arm, Shoulder and Hand Score (QDASH). | Preoperatively, 3 months, 6 months and 12 months postoperatively
  Self-report questionnaire that patients can rate difficulty and interference with daily life on a 5 point Likert scale.

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - MORE Foundation, Phoenix, Arizona
  - Banner Health, Tuscon, Arizona
  - University of Iowa, Iowa City, Iowa
  - Duke University, Durham, North Carolina
  - West Virginia University, Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: No